CLINICAL TRIAL: NCT02180373
Title: Understanding Peripheral Restenosis: Genomic and Proteomic Determinants of Vascular Intervention
Brief Title: PREDICT-PVI Understanding Peripheral Restenosis: Genomic and Proteomic Determinants of Vascular Intervention
Status: Completed | Type: Observational
Sponsor: Vascular Cures (Other)
Responsible Party: Sponsor
Other Study IDs: VCures
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2021-10-05 (Actual); Status verified 2021-10

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Whole blood from 3 timepoints plus 1 tube of plasma; for vein graft bypass arm, otherwise discarded vein tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- vein graft bypass: patients who have had peripheral bypass
- SFA stent: Patients who have had SFA stenting

SUMMARY:
The overall goal of this multicenter collaborative research study is to identify genetic, proteomic, and/or lipidic (lipidomic) biomarkers associated with the outcomes of lower extremity revascularization in patients with advanced peripheral artery disease (PAD).

DETAILED DESCRIPTION:
Vascular surgeons at 10-15 centers will ultimately be involved. Patients who are already undergoing physician-specified intervention and follow up, and meet enrollment criteria, will participate in the study. The PREDICT study includes two independent arms to assess restenosis - peripheral vein graft (VG) bypass surgery and endovascular (angioplasty and superficial femoral artery (SFA) stenting). In broad outline, approximately 1,000 patients will be enrolled for each arm, with clinical follow-up out to two years. Demographic, clinical, and procedural data will be collected at baseline. Clinical and imaging data will be obtained over the follow up period in accordance with standard post-procedural surveillance practices (1, 3, 6, 12, 18, 24 months). Blood samples will be obtained for genomic DNA and plasma biomarkers at 3 time points - baseline, 1 month and 6 months. The baseline samples will provide key information about patients with advanced PAD, often correlated with significant coronary disease.

Data is entered by clinical coordinators into electronic case report forms in the Remedy Informatics database controlled by Vascular Cures. No PHI is included. Paper copies are maintained at the site. Registry data elements were developed with the study PI at University of California at San Francisco (UCSF). The Vascular Cures project manager reviews the database on a monthly basis to insure that case report forms (CRFs) are being completed appropriately and manage the data. Minor data omissions will be ignored; coordinators will be asked to re-submit for any major omissions. Site coordinators are responsible for managing all activities related to patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years.
2. Provision of written informed consent for biospecimen storage, broad genetic and proteomic analysis of tissues, without restrictions, and correlation with clinical outcome data.
3. Willingness to undergo all study collection procedures and sample analyses

   . VG BYPASS COHORT

1. Patient requires placement of an infrainguinal vein bypass graft for the treatment of chronic peripheral artery occlusive disease (PAD). Disabling claudication or critical limb ischemia are acceptable indications.

2. Adequate vein conduit (saphenous vein or alternative vein/spliced vein grafts) for bypass available based on preoperative surgical and/or ultrasound assessment.

SFA COHORT:

1. Patient requires placement of a superficial femoral artery stent for the treatment of chronic peripheral artery occlusive disease (PAD). Disabling claudication or critical limb ischemia are acceptable indications.
2. TransAtlantic Intersociety Consensus (TASC) A-C lesions (must be >70% by visual estimate) amenable to bare metal or drug-eluting stent placement. Stent manufacturer is at the discretion of the treating physician; stents to be used must be commercially available and, if drug-eluting, FDA-approved for SFA use .
3. Must have at least one patent outflow vessel to the foot.

Exclusion Criteria:

1. Anticipated life expectancy less than 2 years.
2. Undergoing active treatment for advanced malignancy (e.g. metastatic disease).
3. On immunosuppressive therapy for solid organ transplant or other indications.
4. Known or suspected hypercoagulable state.
5. Unable or unwilling to be compliant with the follow-up assessments.

VG BYPASS COHORT

1. Use of any non-autogenous conduit or revision of a pre-existing graft.
2. Bypass performed for other than chronic atherosclerotic occlusive disease (e.g. arteritis, aneurysm, acute limb ischemia or trauma).
3. Combined endovascular intervention during same procedure (i.e. hybrid procedure) except for treatment of ipsilateral TASC A/B iliac disease.

SFA STENT COHORT

1. Stent placement performed for other than chronic atherosclerotic occlusive disease (e.g. arteritis, aneurysm, acute limb ischemia, or trauma).
2. TASC D disease (total SFA occlusion or occlusion with severe calcification not amenable to stent placement).
3. Previous SFA stent placement.
4. Use of stent graft.
5. Lesions requiring stent placement > 1cm below the tibial plateau.
6. Known or suspected allergy to nickel.
7. Pregnancy.

   -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced peripheral artery disease already undergoing treatment by participating vascular surgeons, who are either having vein graft (VG) bypass or superficial femoral artery (SFA) stenting. These procedures are unrelated to this study. Enrollment is at the discretion of the participating vascular surgeon in addition to meeting inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-12; Primary Completion 2017-07-28 (Actual); Study Completion 2017-07-28 (Actual)

PRIMARY OUTCOMES:
Revascularization required | 2 years
  observation is to identify biomarkers of vascular healing

CONTACTS AND LOCATIONS:
Overall Officials: Michael S Conte, MD, Principal Investigator — University of California, San Francisco
Locations (4):
- United States (4):
  - UCSF, San Francisco, California
  - University of Florida, Gainesville, Florida
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Puget Sound VA, Seattle, Washington